CLINICAL TRIAL: NCT01594671
Title: Prevention of Postoperative Blood Loss: Randomised Multicentre Parallel Clinical Trial That Assess the Topical and Intravenous Tranexamic Acid in Surgical Patients With a Total Knee Arthroplasty.
Brief Title: Tranexamic Acid for Unilateral Total Knee Arthroplasty
Acronym: TRANEXTOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IIBSP-ATR-2010-23
Record Dates: First submitted 2012-05-03; First posted 2012-05-09 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Blood Loss
Keywords: primary knee arthroplasty; tranexamic acid; topical
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tranexamic acid (Experimental): Intravenous Tranexamic Acid Two dosage Tranexamic acid during the surgical intervention: the first dosage 15-30' before the leg ischemia and the second dosage at 60 -90' after the first dosage.
  Each dosage: 2 ampoules of 500mg/5 mL/ampoule Other Name: Amchafibrin
  Interventions: Drug: Tranexamic Acid; Other: haemostasia
- Habitual haemostasia (Active Comparator): The surgical habitual haemostasia.
  Interventions: Other: haemostasia
- Topical Tranexamic acid (Experimental): Topical Tranexamic acid one dose before the closure of the knee joint: a solution containing 1g of tranexamic acid in 50 ml of normal saline (0.9% sodium chloride) applied with a syringe diffuser.
  Interventions: Drug: Tranexamic Acid; Other: haemostasia

INTERVENTIONS:
Drug: Tranexamic Acid — Two dosage during the surgical intervention: the first dosage 15-30' before the leg ischemia and the second dosage at 60 -90' after the first dosage.
  Each dosage: 2 ampoules of 500mg/5 mL/ampoule
  Other Names: Amchafibrin
  Arms: Tranexamic acid
Drug: Tranexamic Acid — One dose before the closure of the knee joint: a solution containing 1g of tranexamic acid in 50 ml of normal saline (0.9% sodium chloride) applied with a syringe diffuser.
  Other Names: Amchafibrin
  Arms: Topical Tranexamic acid
Other: haemostasia — The surgical habitual haemostasia: electrocoagulation of the bleeding tissues

SUMMARY:
Total knee arthroplasty is often associated with excessive postoperative bleeding due to increased fibrinolysis. Hence, the objective of the proposed of this multicentre study is to determine the peri-operative bleeding comparing the application of topical and intravenous tranexamic acid with the habitual surgical haemostasis.

DETAILED DESCRIPTION:
Objectives:

1. Principal: To assess if the topical and intravenous tranexamic acid reduce less or at least than 20% the blood losses with respect to the habitual haemostasia in patients, after unilateral total knee arthroplasty.
2. Secondary: To assess the treatment safety. To perform a cost- analyses.

Methods: Randomized, multicentre, open and parallel clinical trial with three comparative groups: Topical tranexamic acid, Intravenous tranexamic acid and habitual haemostasia. In all patients, a single drainage of 8mm will be inserted in the joint, and it will remain closed during one hour after the closure of the skin.

Nº of participant centres: 2. Random allocation will be centralised in "Hospital de la Santa Creu i Sant Pau".

Main outcome: Total blood loss (mL) in the post-operative period collected by the habitual drain system ).

Secondary outcomes: Total blood loss (mL)and hidden blood calculated by Nadler's formula. Proportion of patients with blood transfusion, complications of surgery wound, haemoglobin pre and post-operative, units of blood transfused, post-operative mortality, days of hospital stay, safety of interventions assessed.Direct cost analysis.

Substudy: Pharmacokinetic study. The first 24 patients included in "Hospital de la Santa Creu i Sant Pau" for tranexamic acid (12 topical- 12 intravenous) to determine:

1. Plasmatic concentrations of tranexamic acid
2. In topical and intravenous tranexamic acid administration determine the absorption rate and drug bioavailability by these routes: maximum plasma concentration, time to reach Cmax, AUC, and half-life.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Total knee arthroplasty
* The patient consent to participate

Exclusion Criteria:

* Antecedent of thromboembolic disease
* Patient with cardiac alterations of the rhythm
* Patients with valvular cardiac prosthesis
* Patients with pro-thrombotic alterations of coagulation
* Treatment with anticonceptive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Total blood loss (mL) | at 24 hours postoperatively
  Blood will be collected by drainages during the first 24 hours after surgery.

SECONDARY OUTCOMES:
Hidden blood loss | From admission to hospital until an average of 5 days postoperative period
  Hidden blood loss will be calculated by Nadler's formula
Wound complications | 5 weeks postoperatively
  We will quantify infections, haematomas and other complications related with surgery
Adverse effect related with the interventions | 5 weeks postoperatively
  Any adverse effects related with tranexamic acid will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Aguilera X, M.D, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Martinez-Zapata MJ, PhD, Study Director — Centro Cochrane Iberoamericano. IIB Sant Pau
Locations (2):
- Spain (2):
  - Hospital de la Esperanza, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona